CLINICAL TRIAL: NCT04166136
Title: Efficacy of the Transition of the Foot Strike Pattern From Rearfoot to Midfoot or Forefoot During Running on Pain and Disability in Cadets With Chronic Musculoskeletal Pain
Brief Title: Efficacy of the Transition of the Foot Strike Pattern on Pain and Disability in Cadets With Musculoskeletal Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the pandemic
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Naval School (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFSP
Record Dates: First submitted 2019-06-01; First posted 2019-11-18 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: musculoskeletal pain; physiotherapy; military; running
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The permanence of the new foot strike pattern will be investigated as mediator of the pain and disability outcomes in the presence of the forefoot / midfoot pattern. It will be assessed by a blind assessor through observation of the participants' running footage using their usual sneakers three months after randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Treatment Group (Active Comparator): This group will perform standard physiotherapeutic treatment performed at the Naval School. This treatment consists of the application of conventional TENS whose parameters are: alternating current, rectangular pulse, pulse duration 100μs, frequency of 100Hz for 12000 seconds. Laser therapy with an energy of 5 J at each point, irradiation area of 1cm², irradiation time of 20 seconds, 30 repetitions and total time of 6000 seconds.
  Interventions: Other: Usual Treatment Group
- Transition from the Rearfoot to the Forefoot and Midfoot (Active Comparator): Participants in this group will perform a training aimed at the transition of foot strike pattern from the rearfoot to the forefoot and midfoot progressively. Initially a ten-minute race will be held at a comfortable warm-up speed. Then the participants in this group will run continuously at the usual treadmill speed for thirty minutes in a 12-week progressive training program. The participants will receive verbal command "Try to touch first with the middle region of the foot on the treadmill". In the last four sessions, feedback will be gradually removed. At the end of each session, participants will be asked a question about the naturalness of running the new foot touch pattern on the ground. A scale from 0 to 10 will be used, where 0 means "very difficult to perform" and 10 indicates "easy" pattern. The perception of pain will also be evaluated with the numerical scale of pain of 11 points (0 to 10), where 0 means "no pain" and 10 "the greatest pain possible".
  Interventions: Other: Transition from the Rearfoot to the Forefoot and Midfoot
- Muscle Strengthening Group (Active Comparator): The participants of this group will perform muscle strengthening exercises for trunk and lower limbs divided into four phases of three weeks each. The total period of the program strength will be 12 weeks. Elastos® elastic bands of weak, medium and strong intensity will be used to provide progression to the exercises. The exercises will be supervised and supervised by two physiotherapists. A Phase 1 will consist of four exercises; a phase 2, phase 3 and phase 4 will consist of five different exercises each one. In addition to the muscle strengthening le strengthening protocol, this group will have free access to the standard physiotherapeutic treatment performed at the Naval School during and after the study.
  Interventions: Other: Muscle Strengthening Group

INTERVENTIONS:
Other: Transition from the Rearfoot to the Forefoot and Midfoot — Participants in this group will perform a training aimed at the transition of foot strike pattern from the rearfoot to the forefoot and midfoot progressively. Initially a ten-minute race will be held at a comfortable warm-up speed. Then the participants in this group will run continuously at the usual treadmill speed for thirty minutes in a 12-week progressive training program. Participants will run shod and barefoot alternately. Each week the barefoot running time increased to 30 minutes.
  Arms: Transition from the Rearfoot to the Forefoot and Midfoot
Other: Usual Treatment Group — This group will perform standard physiotherapeutic treatment performed at the Naval School. This treatment consists of the application of conventional TENS whose parameters are: alternating current, rectangular pulse, pulse duration 100μs, frequency of 100Hz for 12000 seconds. Laser therapy with an energy of 5 J at each point, irradiation area of 1cm², irradiation time of 20 seconds, 30 repetitions and total time of 6000 seconds.
  Arms: Usual Treatment Group
Other: Muscle Strengthening Group — The participants of this group will perform muscle strengthening exercises for trunk and lower limbs divided into four phases of three weeks each. The total period of the program strength will be 12 weeks. Elastos® elastic bands of weak, medium and strong intensity will be used to provide progression to the exercises. The exercises will be supervised and supervised by two physiotherapists. A Phase 1 will consist of four exercises; a phase 2, phase 3 and phase 4 will consist of five different exercises each one. In addition to the muscle strengthening le strengthening protocol, this group will have free access to the standard physiotherapeutic treatment performed at the Naval School during and after the study.
  Arms: Muscle Strengthening Group

SUMMARY:
To investigate the efficacy of the footstrike pattern transition from rearfoot to midfoot / forefoot pattern compared to lower limb muscle strengthening exercises and lumbar spine region on decreasing the intensity of chronic musculoskeletal pain in cadets from Naval School. Methods: A randomized controlled trial with blind evaluator and allocation of participants in three parallel groups will be performed. Participating in the study, 81 cadets of the Naval Academy of Rio de Janeiro, between 18 and 24 years of age with chronic musculoskeletal pain in the lower limbs or in the lumbar region and who have the rearfoot as footstrike pattern. Participants will be randomly assigned into the following groups: (1) footstrike pattern transition from rearfoot to midfoot / forefoot; (2) muscle strengthening of the lower limbs and lower back; and (3) usual treatment group. Primary treatment outcomes will be pain and specific disability measured twelve weeks after randomization. Secondary treatment outcomes will be pain and specific disability measured six and nine months after randomization. An intention-to-treat analysis will be performed using mixed linear models to compare outcomes between groups.

DETAILED DESCRIPTION:
A total of 81 participants will be enrolled in the study, randomized and allocated to one of the following three groups Usual Treatment Group: This group will perform standard physiotherapeutic treatment performed at the Naval School. This treatment consists of the application of conventional TENS whose parameters are: alternating current, rectangular pulse, pulse duration 100μs, frequency of 100Hz for 20 minutes. Laser therapy with an energy of 5 J at each point, irradiation area of 1cm², irradiation time of 20 seconds, 30 repetitions and total time of 10 minutes.

4.4.3 Transition from the Rearfoot to the Forefoot and Midfoot Group: Participants in this group will perform a training aimed at the transition of foot strike pattern from the rearfoot to the forefoot and midfoot progressively. Initially a ten-minute race will be held at a comfortable warm-up speed. Then the participants in this group will run continuously at the usual treadmill speed for thirty minutes in a 12-week progressive training program. See below: Week 1: 1min of barefoot running + 29 min of shod running Week 2: 2min of barefoot running + 28 min of shod running Week 3: 3min of barefoot running + 27 min of shod running Week 4: 5min of barefoot running + 25 min of shod running Week 5: 1min of barefoot running + 3 min of shod running (repeat 7 times) + 2 finals minuntes shod running Week 6: 1min of barefoot running +3 min of shod running (repeat 10 times) Week 7: 1min of barefoot running +1 min of shod running (repeat 15 times) Week 8: 10 min continuous of barefoot running + 20 min continuous of shod running Week 9: 15 min continuous of barefoot running + 15 min continuous of shod running Week 10: 20 min continuous of barefoot running + 10 min continuous of shod running Week 11: 25 min continuous of barefoot running + 5 min continuous of shod running Week 12: 30 min continuous of barefoot running Participants will receive verbal command "Avoid touching first with heel on the treadmill" and "Try to touch first with the middle region of the foot on the treadmill". If necessary, the investigator will provide additional feedback with verbal details about the foot strike pattern. During the first eight sessions continuous feedback will be given. In the last four sessions, feedback will be gradually removed. At the end of each session, participants will be asked a question about the naturalness of running the new foot touch pattern on the ground. A scale from 0 to 10 will be used, where 0 means "very difficult to perform / unnatural standard" and 10 indicates "easy / natural" pattern. The perception of pain will also be evaluated with the numerical scale of pain of 11 points (0 to 10), where 0 means "no pain" and 10 "the greatest pain possible". Weekly participants will receive visual feedback through slow-motion footage of their footfall during the race, along with investigator guidance on the new tread pattern. In addition to the treadmill transition protocol, this group will have free access to the standard physiotherapeutic treatment performed at the Naval School during and after the study.

Muscle Strengthening Group: The participants of this group will perform muscle strengthening exercises for trunk and lower limbs divided into four phases of three weeks each, following the protocol adapted from Esculier et al. (Esculier et al., 2017) The total period of the program strength will be 12 weeks. Elastos® elastic bands of weak, medium and strong intensity will be used to provide progression to the exercises. The exercises will be supervised by two investigators.

1. A Phase 1 will consist of four exercises:

   I. Participant lying sideways, raise the upper leg while lightly pushing it back. Hold position. The exercise should be performed on both sides of the body 2 times a week. In the first week, 2 sets with 10 repetitions and permanence time of 5 seconds, with progression in the following weeks to 15 repetitions of 10 seconds. An elastic band will be worn around the legs at the ankles.

   II. Participant lying sideways, knees bent, raise the upper knee. The pelvis should remain stable, both feet together. The exercise should be performed on both sides of the body 2 times a week. In the first week, 2 sets with 10 repetitions and stay time of 5 seconds, with progression in the following weeks to 15 repetitions of 10 seconds. An elastic band will be worn around the legs at the knees.

   III. Participant lying on the back, knees bent, raise the pelvis and hold the bridge position. Extend one of the knees (one-sided bridge). The pelvis should remain elevated. The exercise should be performed with both legs 2 times a week. In the first week, 2 sets with 10 repetitions and 5 seconds permanence time, with progression in the following weeks for 15 repetitions of 10 seconds IV. Participant looking at the mirror, step up the step slowly. Step down slowly with the same leg keeping the alignment of the knee and pelvis. The exercise should be performed with the 2 legs, 2 times a week. In the first week, 2 sets with 10 repetitions in the step with 10 cm in height, with progression in the following weeks for 15 repetitions and the height of the step to 20 centimeters.
2. Phase 2 will consist of five exercises:

   V. Participant stand, with elastic band around the knees, squat while keeping the knees in line with the feet (squatting). Do not allow the tip of the knees to move in front of the feet. The exercise should be performed twice a week. In the first week, 2 sets with 10 repetitions and 5 seconds permanence time, with progression in the following weeks for 15 repetitions of 10 seconds.

   VI. Participant looking at the mirror, step down slowly. Step up again with the same leg keeping the focus on aligning the knees. The exercise should be performed with both legs 2 times a week. In the first week, 3 sets with 10 repetitions in the step with 10 cm in height. with progression in the following weeks for 15 repetitions and the height of the step to 20 centimeters.

   VII. Participant with the elastic band around the ankles, push in 3 different directions using the hip musculature. The exercise should be performed with both legs, 2 times a week, 10 repetitions per direction and in 3 directions. The elastic tension is increased as needed.

   VIII. Participant holding the body up using elbows and forearms, raise the pelvis and keep the back straight (plank). Hold this position. The exercise should be performed twice a week. In the first week, 5 replicates with a 10 second residence time, with progression in the following weeks to 10 repetitions of 10 seconds.

   IX. Participant on the side, supporting the body using elbow and forearm, raise the pelvis and keep the back straight (lateral board). Hold this position. Exercise should be performed on both sides. The exercise should be performed twice a week. In the first week, 5 replicates with a 10 second residence time, with progression in the following weeks to 10 repetitions of 10 seconds.
3. Phase 3 will consist of five exercises:

   X. Participant standing on one leg, squat, hold the knee toward the foot (one-sided squat). Hold this position. The exercise should be performed with both legs 2 times a week. In the first week, 2 sets with 10 repetitions and 5 seconds permanence time, with progression in the following weeks for 15 repetitions of 10 seconds.

   XI. Participant looking at the mirror, on a step and with an elastic pulling the knee inward step down and step up slowly. The exercise should be performed with both legs 2 times a week. In the first week, 2 sets with 10 repetitions in the step with 10 cm in height, with progression in the following weeks for 15 repetitions in a step of 20 centimeters.

   XII. Participant standing on one leg, perform the squat while rotating the trunk. Touch the outside of the foot using the opposite hand. Stay in that position. Return to the starting position by turning the hip. The exercise should be performed with both legs 2 times a week. In the first week, 2 sets with 10 repetitions and 5 seconds permanence time, with progression in the following weeks for 2 sets with 15 repetitions and 10 seconds of permanence.

   XIII. Participant holding the body up using elbows and forearms, elevate the pelvis. Remove one foot from the ground while remaining with the knee extended. Hold this position. The exercise should be performed with both legs 2 times a week. In the first week, 2 repetitions with 10 second permanence time in each leg, with progression to 5 repetitions of 10 seconds in each leg.

   XIV. Participant on the side, supporting the body using elbow and forearm, raise the pelvis, keep the back straight (unilateral board) while raising the upper leg. Hold this position. Exercise should be performed on both sides. The exercise should be performed twice a week. In the first week, 5 repetitions and 10 second permanence time with progression in the following weeks for 10 repetitions and 10 second permanence time.
4. Phase 4 will consist of five exercises:

XV. Participant looking at the mirror, with an elastic pulling the knee inward perform a squat while maintaining the alignment of the knee. The other leg stays forward, with the foot off the ground. Hold this position. The exercise should be performed with both legs 2 times a week. In the first week, 2 sets with 10 repetitions and 5 seconds permanence time, with progression in the following weeks for 15 repetitions of 10 seconds.

XVI. Participant looking at the mirror, on top of a step and with a stronger elastic than the one used in exercise XI pulling the knee inward, step down and step up slowly. The exercise should be performed with both legs 2 times a week. In the first week, 3 sets with 10 repetitions in the step with 10 cm in height, with progression in the following weeks for 15 repetitions in a step of 20 centimeters.

XVII. Participant standing on one leg and looking at the mirror, jump off the step with one leg and land smoothly in the squatting position. Be sure to keep good control of the knee and pelvis. An elastic strap pulling the support knee inward can be used to increase the difficulty. The exercise should be performed with both legs 2 times a week. In the first week, 2 sets with 10 repetitions in the step with 10 cm in height, with progression in the following weeks for 15 repetitions in a step of 20 centimeters.

XVIII. Participant holding the body up using elbows and forearms resting on flexible balance discs, elevate the pelvis. Remove one foot from the ground while remaining with the knee extended. Hold this position. The exercise should be performed with both legs 2 times a week. In the first week, 2 repetitions with 10 second permanence time in each leg, with progression to 5 repetitions of 10 seconds in each leg.

XIX. Participant on the side, supporting the body using elbow and forearm supported on a flexible balancing disc, raise the pelvis, keep the back straight (unilateral board) while raising the upper leg. Hold this position. Exercise should be performed on both sides. The exercise should be performed twice a week. In the first week, 5 repetitions and 10 second permanence time with progression in the following weeks for 10 10 second repetitions.

In addition to the muscle strengthening protocol, this group will have free access to the standard physiotherapeutic treatment performed at the Naval School during and after the study.

ELIGIBILITY:
Inclusion Criteria:

1. chronic musculoskeletal pain in the lower limbs and / or non-specific chronic low back pain that is related to running ("persistent pain" will be considered "chronic" for more than three months). Information on pain will be based on a self-completion questionnaire;
2. rearfoot as a foot strike pattern;
3. present at least one run-related limitation on the Specific Functional Scale of the Patient (EFEP);
4. practice running 2 to 5 times a week.

Exclusion Criteria:

1. have undergone a surgical procedure in the lower limbs and / or the lower back in the last six months;
2. have performed invasive procedures for pain relief in the last three months; do not present a history of acute trauma such as fractures in the last six months, infection, signs of radiculopathy, compression of the marrow or equine tail.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity: Brazilian version of the Numerical Pain Scale | Three months after randomization
  Pain intensity will be measured using the Brazilian version of the Numerical Pain Scale,whose ranges from 0 to 10, where 0 represents "no pain" and 10 represents "the worst possible pain" based on the last seven days.
Specific disability | Three months after randomization
  Specific disability through the Patient Specific Functional Scale. At this scale, the participant should report three activities whose achievements are being hampered by pain. Participant should note the difficulty on a scale of 0 to 10, where 0 means "unable to perform activity" and 10 means "able to perform the activity as you did before the injury."

SECONDARY OUTCOMES:
Weekly running mileage | Three months after randomization
  Weekly running mileage will be obtained through a self-completion questionnaire in which participants will answer the following question: "How many kilometers do you run per week?".
Weekly running mileage | Six months after randomization
  Weekly running mileage will be obtained through a self-completion questionnaire in which participants will answer the following question: "How many kilometers do you run per week?".
Pain intensity: Brazilian version of the Numerical Pain Scale | Six months after randomisation
  Pain intensity will be measured using the Brazilian version of the Numerical Pain Scale,whose ranges from 0 to 10, where 0 represents "no pain" and 10 represents "the worst possible pain" based on the last seven days.
Specific disability | Six months after randomisation
  Specific disability through the Patient Specific Functional Scale. At this scale, the participant should report three activities whose achievements are being hampered by pain. Participant should note the difficulty on a scale of 0 to 10, where 0 means "unable to perform activity" and 10 means "able to perform the activity as you did before the injury."

CONTACTS AND LOCATIONS:
Overall Officials: Ney Meziat, PhD, Principal Investigator — Centro Universitario Augusto Motta, UNISUAM
Locations (2):
- Brazil (2):
  - UNISUAM, Rio de Janeiro, Rio de Janeiro
  - Centro Universitário Augusto Motta, Rio de Janeiro

REFERENCES:
- [Background] Almeida MO, Davis IS, Lopes AD. Biomechanical Differences of Foot-Strike Patterns During Running: A Systematic Review With Meta-analysis. J Orthop Sports Phys Ther. 2015 Oct;45(10):738-55. doi: 10.2519/jospt.2015.6019. Epub 2015 Aug 24. PMID 26304644
- [Background] Barton CJ, Levinger P, Crossley KM, Webster KE, Menz HB. The relationship between rearfoot, tibial and hip kinematics in individuals with patellofemoral pain syndrome. Clin Biomech (Bristol). 2012 Aug;27(7):702-5. doi: 10.1016/j.clinbiomech.2012.02.007. Epub 2012 Mar 20. PMID 22436492
- [Background] Boling M, Padua D, Marshall S, Guskiewicz K, Pyne S, Beutler A. Gender differences in the incidence and prevalence of patellofemoral pain syndrome. Scand J Med Sci Sports. 2010 Oct;20(5):725-30. doi: 10.1111/j.1600-0838.2009.00996.x. PMID 19765240
- [Background] Bullock SH, Jones BH, Gilchrist J, Marshall SW. Prevention of physical training-related injuries recommendations for the military and other active populations based on expedited systematic reviews. Am J Prev Med. 2010 Jan;38(1 Suppl):S156-81. doi: 10.1016/j.amepre.2009.10.023. PMID 20117590
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Crofford LJ. Chronic Pain: Where the Body Meets the Brain. Trans Am Clin Climatol Assoc. 2015;126:167-83. PMID 26330672
- [Background] de Almeida MO, Saragiotto BT, Yamato TP, Lopes AD. Is the rearfoot pattern the most frequently foot strike pattern among recreational shod distance runners? Phys Ther Sport. 2015 Feb;16(1):29-33. doi: 10.1016/j.ptsp.2014.02.005. Epub 2014 Feb 26. PMID 24894762
- [Background] Diebal AR, Gregory R, Alitz C, Gerber JP. Forefoot running improves pain and disability associated with chronic exertional compartment syndrome. Am J Sports Med. 2012 May;40(5):1060-7. doi: 10.1177/0363546512439182. Epub 2012 Mar 16. PMID 22427621
- [Background] Esculier JF, Bouyer LJ, Dubois B, Fremont P, Moore L, McFadyen B, Roy JS. Is combining gait retraining or an exercise programme with education better than education alone in treating runners with patellofemoral pain?A randomised clinical trial. Br J Sports Med. 2018 May;52(10):659-666. doi: 10.1136/bjsports-2016-096988. Epub 2017 May 5. PMID 28476901
- [Background] Esculier JF, Silvini T, Bouyer LJ, Roy JS. Video-based assessment of foot strike pattern and step rate is valid and reliable in runners with patellofemoral pain. Phys Ther Sport. 2018 Jan;29:108-112. doi: 10.1016/j.ptsp.2016.11.003. Epub 2016 Nov 23. PMID 28666810
- [Background] Hauret KG, Jones BH, Bullock SH, Canham-Chervak M, Canada S. Musculoskeletal injuries description of an under-recognized injury problem among military personnel. Am J Prev Med. 2010 Jan;38(1 Suppl):S61-70. doi: 10.1016/j.amepre.2009.10.021. PMID 20117601
- [Background] Hespanhol Junior LC, Pena Costa LO, Lopes AD. Previous injuries and some training characteristics predict running-related injuries in recreational runners: a prospective cohort study. J Physiother. 2013 Dec;59(4):263-9. doi: 10.1016/S1836-9553(13)70203-0. PMID 24287220
- [Background] Knapik JJ, Graham B, Cobbs J, Thompson D, Steelman R, Jones BH. A prospective investigation of injury incidence and injury risk factors among Army recruits in military police training. BMC Musculoskelet Disord. 2013 Jan 17;14:32. doi: 10.1186/1471-2474-14-32. PMID 23327563
- [Background] Louw M, Deary C. The biomechanical variables involved in the aetiology of iliotibial band syndrome in distance runners - A systematic review of the literature. Phys Ther Sport. 2014 Feb;15(1):64-75. doi: 10.1016/j.ptsp.2013.07.002. Epub 2013 Aug 16. PMID 23954385
- [Background] Nunns M, House C, Fallowfield J, Allsopp A, Dixon S. Biomechanical characteristics of barefoot footstrike modalities. J Biomech. 2013 Oct 18;46(15):2603-10. doi: 10.1016/j.jbiomech.2013.08.009. Epub 2013 Aug 27. PMID 24054331
- [Background] Nye NS, Pawlak MT, Webber BJ, Tchandja JN, Milner MR. Description and Rate of Musculoskeletal Injuries in Air Force Basic Military Trainees, 2012-2014. J Athl Train. 2016 Nov;51(11):858-865. doi: 10.4085/1062-6050-51.10.10. PMID 28068163
- [Background] Roper JL, Harding EM, Doerfler D, Dexter JG, Kravitz L, Dufek JS, Mermier CM. The effects of gait retraining in runners with patellofemoral pain: A randomized trial. Clin Biomech (Bristol). 2016 Jun;35:14-22. doi: 10.1016/j.clinbiomech.2016.03.010. Epub 2016 Apr 7. PMID 27111879
- [Background] Salsich GB, Graci V, Maxam DE. The effects of movement pattern modification on lower extremity kinematics and pain in women with patellofemoral pain. J Orthop Sports Phys Ther. 2012 Dec;42(12):1017-24. doi: 10.2519/jospt.2012.4231. Epub 2012 Sep 5. PMID 22960572
- [Background] Santuz A, Ekizos A, Janshen L, Baltzopoulos V, Arampatzis A. The Influence of Footwear on the Modular Organization of Running. Front Physiol. 2017 Nov 22;8:958. doi: 10.3389/fphys.2017.00958. eCollection 2017. PMID 29213246

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT04166136/SAP_001.pdf
  • Informed Consent Form (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT04166136/ICF_000.pdf